CLINICAL TRIAL: NCT00215215
Title: Post Marketing Study; Randomized, Parallel-Group Comparison of Treatment With Pharmacotherapy or Adjunctive Vagus Nerve Stimulation Therapy for Pharmacoresistant Partial Seizures: A Large Simple Effectiveness Trial
Brief Title: Effectiveness Study Comparing Treatment With Drug(s) or Adjunctive VNS Therapy for Pharmacoresistant Partial Seizures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Cyberonics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-20
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2006-02

CONDITIONS: Epilepsies, Partial
Keywords: Vagus Nerve Stimulation Therapy; Epilepsies, Partial; Seizures; Antiepileptic Drugs; Refractory Partial Seizures
MeSH Terms: conditions — Epilepsies, Partial; Seizures

INTERVENTIONS:
Device: Vagus Nerve Stimulation Therapy

SUMMARY:
To compare outcomes over 12 months of treatment with antiepileptic drugs (AEDs) alone or vagus nerve stimulation (VNS) therapy plus AEDs in patients who have partial seizures refractory to at least two, but not more than five, AEDs.

DETAILED DESCRIPTION:
Published data suggest that patients who continue to experience seizures after trials of two or three AEDs are unlikely to become seizure-free with further attempts at pharmacotherapy. Such patients may experience poor quality of life and functional outcomes from continuing seizures and the adverse effects associated with further attempts at pharmacotherapy. VNS is a non-pharmacologic treatment for epilepsy with well-established effectiveness as an adjunctive treatment (to AEDs) for partial seizures refractory to AEDs, but there are no randomized clinical trials comparing the effectiveness of adjunctive VNS therapy with further pharmacotherapy alone in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of partial seizures with onset before age 50, and the patient's prior electroencephalography and magnetic resonance imaging studies are consistent with the diagnosis of partial seizures.
* Patient has at least 4 complex partial seizures, but less than 25 seizures (any type), per month during the 3 months preceding randomization; for the 8 weeks preceding randomization, the seizure frequency should be confirmed from a patient diary.
* Patient has not had an adequate response to an adequate dosage of -- or was intolerant to -- a minimum of 2 different AEDs.
* Patient has (in the investigator's judgment) sufficient impairment from his/her epilepsy and/or epilepsy treatment that the potential benefits/risks of VNS therapy are warranted.
* Patient must currently be receiving at least one AED, but not more than three AEDs, in a stable dosage regimen for at least one month before randomization.
* Patient must be 12 years of age or older.
* Patient must be able to provide reliable seizure counts and to complete the evaluations specified in the study procedures flow chart.
* Patient must provide written informed consent, or legal guardian must give written permission and the minor provide written assent.

Exclusion Criteria:

* Patient has a history (lifetime) of having received more than 5 different AEDs.
* Patient has had a bilateral or left cervical vagotomy.
* Patient currently uses, or is expected to use during the study, short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy.
* A VNS Therapy System implant would (in the investigator's judgment) pose an unacceptable surgical or medical risk for the patient.
* Patient is expected to require full body magnetic resonance imaging during the clinical study.
* Patient has had a previous VNS Therapy System implant.
* Patient has a previous neuroimaging study that demonstrates mesial temporal sclerosis, cortical dysplasia, or a suspected brain tumor.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360
Dates: Start 2005-02; Study Completion 2007-11

PRIMARY OUTCOMES:
*Quality of Life in Epilepsy Questionnaire (QOLIE)
at baseline, Week 26 and Week 52.
*Patients will be asked to keep a daily record of their seizures in a seizure diary supplied by the investigational sites.

SECONDARY OUTCOMES:
The QOLIE at baseline, Week 26 and Week 52.
*Percentage Change in Seizure-Related Disability Assessment Scale (SERDAS)at baseline and Week 52 for each patient.
*Percentage Change in Hospital Anxiety and Depression Scale (HAD)at baseline and Week 52 for each patient.
*Over the course of the study, AED medications will be assessed.
*Patient Satisfaction Survey will be performed at Week 52.

CONTACTS AND LOCATIONS:
Overall Officials: Carol C Base, RN, MS, Study Director — Cyberonics, Inc.
Locations (23):
- United States (23):
  - Bronislav Shafran, M.D., P.C., Phoenix, Arizona
  - Xenoscience, Phoenix, Arizona
  - Dedicated Clinical Research, Inc., Sun City, Arizona
  - USC Comprehensive Epilepsy Center, Los Angeles, California
  - Certified Clinical Research, Roseville, California
  - Pediatric Diagnostic Center, Ventura, California
  - University of Florida, Department of Neurology, Gainesville, Florida
  - Neurology Associates, P.A., Maitland, Florida
  - Child Neurology Center of Northwest Florida, Pensacola, Florida
  - Pediatric Neurology of Idaho, Boise, Idaho
  - Freeport Health Network, Department of Neurology, Freeport, Illinois
  - Wayne State University School of Medicine, Department of Neurology, Detroit, Michigan
  - Weill-Cornell Medical College, N.Y. Presbyterian Hospital, Comprehensive Epilepsy Center, New York, New York
  - William Huffstutter, M.D., Asheville, North Carolina
  - Medford Neurological and Spine Clinic, Medford, Oregon
  - Neurology and Sleep Medicine, Bethlehem, Pennsylvania
  - Mid-South Physicians Group, P.L.L.C., Germantown, Tennessee
  - Hermann Hospital, UT Comprehensive Epilepsy Center, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Texas Association of Pediatric Neurology, San Antonio, Texas
  - Pivotal Research Centers, Midvale, Utah
  - Pharmaceutical Research Organization, South Ogden, Utah
  - Regional Epilepsy Center Saint Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Schachter SC. Vagus nerve stimulation therapy summary: five years after FDA approval. Neurology. 2002 Sep 24;59(6 Suppl 4):S15-20. doi: 10.1212/wnl.59.6_suppl_4.s15. PMID 12270963
- [Background] Renfroe JB, Wheless JW. Earlier use of adjunctive vagus nerve stimulation therapy for refractory epilepsy. Neurology. 2002 Sep 24;59(6 Suppl 4):S26-30. doi: 10.1212/wnl.59.6_suppl_4.s26. PMID 12270965
- [Background] Fisher RS, Handforth A. Reassessment: vagus nerve stimulation for epilepsy [RETIRED]: a report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Neurology. 1999 Sep 11;53(4):666-9. doi: 10.1212/wnl.53.4.666. No abstract available. PMID 10489023
- [Background] Heck C, Helmers SL, DeGiorgio CM. Vagus nerve stimulation therapy, epilepsy, and device parameters: scientific basis and recommendations for use. Neurology. 2002 Sep 24;59(6 Suppl 4):S31-7. doi: 10.1212/wnl.59.6_suppl_4.s31. PMID 12270966